CLINICAL TRIAL: NCT01104532
Title: A Phase 1, Open Label, Randomized, Crossover, Drug Interaction Study of the Pharmacokinetics of ASP1941 and Sitagliptin After Separate and Concomitant Administration to Healthy Adult Subjects
Brief Title: A Study to Characterize the Effect on the Pharmacokinetics of ASP1941 and Sitagliptin When Given Together to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sr. Manager Clinical Trials Registry, Astellas Pharma Global Development
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1941-CL-0066
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Healthy; Pharmacokinetics of ASP1941
Keywords: ASP1941; Januvia; sitagliptin
MeSH Terms: interventions — ipragliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dosing Regimen 1 (Experimental)
  Interventions: Drug: ASP1941; Drug: sitagliptin
- Dosing Regimen 2 (Experimental)
  Interventions: Drug: ASP1941; Drug: sitagliptin
- Dosing Regimen 3 (Experimental)
  Interventions: Drug: ASP1941; Drug: sitagliptin
- Dosing Regimen 4 (Experimental)
  Interventions: Drug: ASP1941; Drug: sitagliptin

INTERVENTIONS:
Drug: ASP1941 — oral tablet
Drug: sitagliptin — oral tablet
  Other Names: Januvia

SUMMARY:
The purpose of the study is to evaluate pharmacokinetics, pharmacodynamics and safety following the administration of ASP1941 and sitagliptin in single and multiple doses.

DETAILED DESCRIPTION:
All subjects will be enrolled at one center and confined to the unit for up to 17 days. Subjects will be dosed in the fasting state in one of the four groups.

ELIGIBILITY:
Inclusion Criteria:

* The subject weighs at least 50 kg, and has a body mass index (BMI) of 18 to 32 kg/m2 inclusive
* The subject's 12-lead electrocardiogram (ECG) results are normal
* The female subject must be at least two years postmenopausal, surgically sterile or practicing effective birth control and not pregnant or lactating
* The male or female subject agrees to practice highly effective birth control from Screening until 7 days post last dose

Exclusion Criteria:

* The subject has a history or evidence of any clinically significant cardiovascular, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy (excluding non-melanoma skin cancer)
* The subject has evidence of renal insufficiency (serum creatinine ≥ 1.5 in men and ≥ 1.3 in women)
* The subject has a history of cholelithiasis or acute pancreatitis
* The subject has any condition possibly affecting drug absorption (e.g., gastrectomy)
* The subject has history of consuming more than 14 units of alcoholic beverages per week within last 6 months or has a history of alcoholism or drug/chemical/substance abuse within past 2 years or the subject tests positive for alcohol or drugs of abuse
* The subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic check-in
* The subject has a supine mean systolic blood pressure <90 or >160 mm/Hg and a mean diastolic blood pressure <50 or >90, or pulse rate higher than 100 beats per min (bpm)
* The subject has a 12-lead ECG demonstrating QTcF >470 msec (female) or >450 msec (male)
* The subject is known positive for human immunodeficiency virus (HIV) antibody
* The subject has a positive test for tuberculosis (TB), hepatitis C antibody, or positive for hepatitis B surface antigen (HGsAg)
* The subject has used prescription or non-prescription drugs within 14 days or 5 half-lives (whichever is longer) or complementary and alternative medicines (CAM) within 14 days prior to study drug administration (excluding oral contraceptives, hormone replacement therapy [HRT], and acetaminophen)
* The subject has been vaccinated within the last 7 days
* The subject has had any significant blood loss, donated one unit (450 mL) or blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables assessment through analysis of blood samples | Day 1 to Day 15

SECONDARY OUTCOMES:
Pharmacodynamic variables assessment through analysis of blood and urine samples | Day -1 and up to Day 11
Safety assessed by recording of adverse events, laboratory assessments, electrocardiograms (ECGs), vital signs and physical examinations | Day 1 through scheduled group check out (Day 11 and up to Day 15) or early termination.

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- Miami, Florida, United States